CLINICAL TRIAL: NCT05227781
Title: 8 Weeks of L-Citrulline Supplementation to Improve Low-intensity Resistance Exercise Training Vascular Adaptations in Postmenopausal Women With Hypertension
Brief Title: 8 Weeks of L-CIT Supplementation and LIRET on Vascular Function in Hypertensive Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Arturo Figueroa, Principal Investigator, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2018-463
Record Dates: First submitted 2021-12-10; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Hypertension; Menopause
Keywords: Endothelial Function; Arterial Stiffness; Muscle Function
MeSH Terms: conditions — Hypertension | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Double-blind (subject, investigator), randomized, parallel, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind, randomized, parallel, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Citrulline (Experimental): L-Citrulline: 10 grams/day
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Maltodextrin: 10 grams/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — 8 weeks of L-Citrulline supplementation (10 grams/day)
  Arms: L-Citrulline
Dietary Supplement: Placebo — 8 weeks of Placebo (maltodextrin; 10 grams/day)
  Arms: Placebo

SUMMARY:
The overall objective of this project is to bring forth evidence that L-Citrulline (L-CIT) supplementation and low intensity resistance exercise training (LIRET) alone and combined will improve vascular function and muscle fitness (mass, strength, and exercise performance) in postmenopausal women with hypertension. The investigators' central hypothesis is that adjuvant L-CIT supplementation may synergistically enhance vascular (arterial stiffness, BP, muscle oxygenation, blood flow) and muscular (strength, exercise performance) responses to LIRET in postmenopausal women with hypertension by improving endothelial vasodilatory function.

DETAILED DESCRIPTION:
Individuals who are on medications will refrain from use the morning of all laboratory visits. Participants will be asked to bring medications with them, and will be allowed to ingest it after the vascular measurements have been obtained.

There will be a total of 7 laboratory visits. The 1st visit will be approximately 1 hr and 45 minutes. The 2nd and 3rd visit will be approximately 2 hrs. The 4th and 6th visit will total about 2 hrs and 15 minutes and finally, the 5th and 7th visit will total about 1hr and 15 minutes. This means the total participant time for laboratory visits will be approximately 12 hours. In addition to this, the second 4 weeks of the 8 week study period will involve coming to the Kinesiology and Sport Management building at Texas Tech University main campus 3 times per week to perform the low-intensity resistance training intervention. These visits should last no more than 30-45 minutes.

The first 3 visits will be separated by 48-72 hrs. Visits 3 and 4 will be separated by 4 weeks (first 4 weeks of LCIT or Placebo supplementation). Visits 4 and 5 will be separated by 48-72 hours. Visits 5 and 6 will again be separated by 4 weeks (Second 4 weeks of LCIT or Placebo supplementation with the addition of Low-intensity resistance exercise in both groups).

Approximately 12 hours total for each of the 7 laboratory visits, as well as 30-45 minutes 3 times per week during the last 4 weeks of the 8 week study.

Using a parallel placebo-controlled design, postmenopausal women with elevated blood pressure or hypertension will be randomized to receive L-CIT supplementation (10g/day) alone for 4 weeks, followed by 4 weeks of L-CIT supplementation in combination with low-intensity resistance training or placebo (maltodextrin) alone for 4 weeks, followed by 4 weeks of placebo in combination with low-intensity resistance training.

Differences between conditions (Citrulline vs Placebo) will be analyzed with independent samples t-test. Two-way ANOVA with repeated measures with Bonferroni adjustments will be used to analyze group (CIT vs. PL) by time (baseline, post-supplementation only, supplement + low-intensity resistance exercise training) interactions between the outcome variables. If group-by-time interactions are detected, post-hoc comparisons will be performed via paired or independent t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-75 years
* Resting systolic BP 120-159 mmHg
* Sedentary (< 60 min of exercise/week)
* Body mass index of 18.5-39.9 kg/m2)
* Fasting glucose < 126 mg/dL
* HbA1c < 6.4%.

Exclusion Criteria:

* Body mass index ≥ 40 or < 18.5 kg/m2
* Diagnosed with type 1 or 2 diabetes mellitus
* Cardiovascular diseases
* Systolic blood pressure > 170 mmHg or on more than two anti-hypertensive medication
* Other chronic diseases such as cancer, asthma, glaucoma, thyroid, kidney, liver and pancreatic disease
* Individuals incorporated in a weight loss program and aerobic or resistance training program
* Heavy smokers (> 20 cigarettes per day)
* Heavy drinkers (> 12 alcoholic drinks per week)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial function via brachial artery flow-mediated dilation (effects of L-Citrulline only) | 4 weeks
  Endothelial function will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone using brachial artery flow-mediated dilation. All measurements will be performed using Doppler ultrasound.
Changes in endothelial function via superficial femoral artery flow-mediated dilation (effects of L-Citrulline only) | 4 weeks
  Endothelial function will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone using superficial femoral artery flow-mediated dilation. All measurements will be performed using Doppler ultrasound.
Changes in endothelial function via brachial artery flow-mediated dilation (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, endothelial function will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs using brachial artery flow-mediated dilation. All measurements will be performed using Doppler ultrasound.
Changes in endothelial function via superficial femoral artery flow-mediated dilation (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, endothelial function will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs using superficial femoral artery flow-mediated dilation. All measurements will be performed using Doppler ultrasound.
Changes in arm exercise blood flow (effects of L-Citrulline only) | 4 weeks
  Blood flow will be measured in the brachial artery during low intensity arm exercise. All measurements will be performed using Doppler ultrasound.
Changes in leg exercise blood flow (effects of L-Citrulline only) | 4 weeks
  Blood flow will be measured in the superficial femoral arteries during low intensity leg exercise. All measurements will be performed using Doppler ultrasound.
Changes in arm exercise blood flow (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, blood flow will be measured in the brachial artery during low intensity arm exercise. All measurements will be performed using Doppler ultrasound.
Changes in leg exercise blood flow (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, blood flow will be measured in the superficial femoral artery during low intensity leg exercise. All measurements will be performed using Doppler ultrasound.

SECONDARY OUTCOMES:
Changes in arterial stiffness via arm, leg, and aortic pulse wave velocity (effects of L-Citrulline only) | 4 weeks
  Arterial stiffness will be assessed using pulse wave velocity of the arm (carotid-radial), leg (femoral-ankle), and aorta (carotid-femoral) at baseline and after 4 weeks of L-Citrulline supplementation alone using applanation tonometry.
Changes in arterial stiffness via arm, leg, and aortic pulse wave velocity (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  Arterial stiffness will be assessed using pulse wave velocity of the arms (carotid-radial), legs (femoral-ankle), and aorta (carotid femoral) using applanation tonometry after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Changes in aortic hemodynamics using pulse wave analysis (effects of L-Citrulline only) | 4 weeks
  The speed and reflection pressures, both representing aortic hemodynamic parameters, will be assessed using radial artery pulses and a validated transfer function (AtCor Medical) at baseline and after 4 weeks of L-Citrulline supplementation alone.
Changes in aortic hemodynamics using pulse wave analysis (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  The speed and reflection pressures, both representing aortic hemodynamic parameters, will be assessed using radial artery pulses and a validated transfer function (AtCor Medical) after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Changes in brachial and aortic blood pressure via automated sphygmomanometry (effects of L-Citrulline only) | 4 weeks
  Brachial and aortic blood pressures (systolic and diastolic) will be assessed using an arm cuff at baseline and after 4 weeks of L-Citrulline supplementation alone.
Changes in brachial and aortic blood pressure via automated sphygmomanometry (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  Brachial and aortic blood pressures (systolic and diastolic) will be assessed using an arm cuff after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Changes in muscle strength (effects of L-Citrulline only) | 4 weeks
  Handgrip and leg strength (leg press, leg extension, leg flexion, calf raises) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Changes in muscle strength (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, handgrip and leg strength (leg press, leg extension, leg flexion, calf raises) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs. These 4 exercises are to be of focus during the training sessions (3 days/week, 12 total training sessions).
Quantification of L-Arginine (effects of L-Citrulline only) | 4 weeks
  Serum levels of L-Arginine (nmol/ul) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Quantification of Arginase (effects of L-Citrulline only) | 4 weeks
  Serum levels ofarginase (pg/mL) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Quantification of nitric oxide (effects of L-Citrulline only) | 4 weeks
  Serum levels ofnitric oxide (umol/L) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Quantification of Endothelin-1 (effects of L-Citrulline only) | 4 weeks
  Serum levels of endothelin-1 (pg/mL) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Quantification of L-Ornithine (effects of L-Citrulline only) | 4 weeks
  Serum levels of L-Ornithine (pmol/ul) will be assessed at baseline and after 4 weeks of L-Citrulline supplementation alone.
Quantification of L-Arginine (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, serum levels of L-Arginine (nmol/ul) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Quantification of arginase (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, serum levels of arginase (pg/mL) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Quantification of nitric oxide (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, serum levels of nitric oxide (umol/L) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Quantification of endothelin-1 (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, serum levels of endothelin-1 (pg/mL) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.
Quantification of L-Ornithine (effects of L-Citrulline combined with low-intensity resistance exercise training) | 4 weeks
  After the 4-week assessment, serum levels of L-Ornithine (pmol/ul) will be assessed after 4 additional weeks of L-Citrulline supplementation with combined low-intensity resistance exercise training with the legs.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participants are to be de-identified. Only anthropometric information and data from the outcome variables will be analyzed. All data will be condensed into an SPSS file, which will then be given to Doctoral Students for analysis. This file will be transferred between hard drives, not sent via email. This is done to ensure that all data remains confidential.